CLINICAL TRIAL: NCT05282459
Title: A Phase Ib/II, Single Center, Open-Label, Safety and Efficacy Study to Improve Anemia in Subjects on Enasidenib With Lower Risk Myelodysplastic Syndrome and Non-proliferative Chronic Myelomonocytic Leukemia Without an IDH2 Mutation
Brief Title: Enasidenib in MDS &Non-proliferative Chronic Myelomonocytic Leukemia w/o IDH2 Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB- 62692; HEM0056 (Other: Stanford); NCI-2022-02837 (Other: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Leukemia; Leukemia, Myeloid; Monocytic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Monocytic, Acute | interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enasidenib mesylat (Experimental): Participants will self administer the enasidenib orally everyday.
  Interventions: Drug: Enasidenib mesylat dose escalation

INTERVENTIONS:
Drug: Enasidenib mesylat dose escalation — Subjects will participate dose escalation with a starting dose of 100 mg. Enasidenib will be self administered orally and daily.
  Other Names: (Idhifa, AG 221)

SUMMARY:
This is a phase 1b/2, open-label, single arm study to evaluate if enasidenib is safe and effective in improving anemia and decreasing transfusion needs in subjects diagnosed with lower risk myelodysplastic syndrome (MDS) or nonproliferative chronic myelomonocytic leukemia (CMML) without a mutation in isocitrate dehydrogenase type 2 (IDH2 wildtype). Other objectives include assessment of improvements in platelet production and characterization of the mechanism of action of enasidenib in enhancing endogenous erythropoiesis.

DETAILED DESCRIPTION:
Primary Objective(s)- To determine the efficacy (response rate) of enasidenib in improving anemia and decreasing RBC transfusion dependence.

Secondary Objective(s)- To determine the tolerability, safety and durability of the erythroid response and identify laboratory parameters as clinical markers of response.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of

   * MDS according to WHO/FAB classification that meets IRSS-R classification of low or intermediate risk disease; and a diagnosed as denovo or secondary MDS (MDS-RS eligible if refractory to or declined luspatercept therapy) OR
   * Dysplastic (nonproliferative) CMML with WBC < 13.0/microL)
2. No disease-modifying therapy (HMA, hydrea) within 2 months of starting study
3. Age ≥ 18 years of age
4. ECOG ≤ 3
5. Negative for IDH2 mutation by NGS or multiplex PCR (SNaPshot)
6. Has symptomatic anemia defined as hemoglobin < 10.5 g/dL with any of the following.

   * Tachypnea
   * Shortness of breath
   * Fatigue
   * Malaise
   * Worsening of cardiovascular function
   * Asthenia
   * Dyspnea on exertion
   * Angina
   * Other subject symptoms the subject reports as being associated with being anemic.
7. Stated willingness to comply with all study procedures and availability for the duration of the study
8. Ability to take oral medication and be willing to adhere to the medication regimen.
9. Females of reproductive potential need to either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with highly effective contraception without interruption, 28 days prior to starting enasidenib, during the study therapy, and for 30 days after last dose of enasidenib
10. For males of reproductive potential: agreement to use of condoms
11. Adequate organ function defined as:

    * Hepatic function: total bilirubin <1.5 x ULN (unless attributable to Gilbert's disease), AST or ALT < 3x ULN
    * Renal function: creatinine clearance > 30 mL/minute, calculated by Cockcroft-Gault formula
12. Ability to understand and the willingness to sign the IRB approved informed consent document.
13. Women of childbearing potential must have negative urine or serum pregnancy test

Exclusion Criteria:

1. Use of concurrent other erythropoietic agents (including epoetin, darbepoetin), G-CSF within 30 days of study enrollment
2. Less than 3 months of life expectancy
3. Significant cardiac disease (NYHA Class IV congestive heart failure, or unstable angina or myocardial infarction within the last 6 months
4. Harbor IDH2 somatic mutations by NGS or PCR
5. Pregnant or breast feeding
6. Any uncontrolled bacterial, fungal, viral or other infection.
7. No known HIV+ or active hepatitis B or C infection, defined as positive viral load for HBV or HCV or a positive surface antigen (HBsAg) test for hepatitis B.
8. Have other causes of anemia: deficiencies in iron, B12, folate; nutritional deficiencies related to gastric surgery, anorexia nervosa, excessive zinc supplementation; gastrointestinal bleed. If nutritional deficiencies can be corrected, potential subject can be rescreened and enrolled if nutritionally replete and still meets eligibility criteria.
9. Any other medical history, including laboratory results, deemed by the Principal Investigator likely to interfere with their participation in the study, or to interfere with the interpretation of the results
10. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Clinical Response: Hematological Improvement - Erythroid (HI-E) | 16 weeks
  Clinical response was assessed as the number of participants achieving a hematological improvement - erythroid (HI-E). Participants will be characterized and stratified as nontransfused (NTD), low-transfusion burden (LTB) and high-transfusion burden (HTB), with response defined as follows.
  * NTD = greater than or equal to 2 consecutive Hb measurements, greater than or equal to 1.5 g/dL for a period of minimum 8 week in an observation period of 16 to 24 week compared to the lowest mean of 2 Hb measurements
  * LTB = 0 units of RBC transfusions
  * HTB = greater than or equal to 4 unit or greater than or equal to 50% reduction in RBC transfusions The outcome will be reported as the number of participants that achieve the response, a number without dispersion.
Related Adverse Events | 12 months
  Toxicity will be assessed as the number of related non serious adverse events and related serious adverse events (SAEs) reported for the 12 cycle treatment period plus follow up. The outcome will be reported as numbers without dispersion.
Time to Hematological Improvement - Erythroid (HI-E) | 16 weeks.
  Time to hematological improvement - erythroid (HI-E) will be assessed as the time from first dose of enasidenib to the first observed hemoglobin response. Participants will be characterized and stratified as nontransfused (NTD), low-transfusion burden (LTB) and high-transfusion burden (HTB), with response defined as follows.
  * NTD = greater than or equal to 2 consecutive Hb measurements, greater than or equal to 1.5 g/dL for a period of minimum 8 week in an observation period of 16 to 24 week compared to the lowest mean of 2 Hb measurements
  * LTB = 0 units of RBC transfusions
  * HTB = greater than or equal to 4 unit or greater than or equal to 50% reduction in RBC transfusions The outcome will be reported as the number of participants that achieve the response, a number without dispersion.
Duration of Hematological Improvement - Erythroid (HI-E) | 16 weeks.
  Duration of Hematological Improvement - Erythroid (HI-E) will be assessed as the time from recorded response to loss of response. Participants will be characterized and stratified as nontransfused (NTD), low-transfusion burden (LTB) and high-transfusion burden (HTB), with response defined as follows.
  * NTD = greater than or equal to 2 consecutive Hb measurements, greater than or equal to 1.5 g/dL for a period of minimum 8 week in an observation period of 16 to 24 week compared to the lowest mean of 2 Hb measurements
  * LTB = 0 units of RBC transfusions
  * HTB = greater than or equal to 4 unit or greater than or equal to 50% reduction in RBC transfusions The outcome will be reported as the number of participants that achieve the response, a number without dispersion.
Clinical Response: Hematological Improvement - Platelets (HI-P) | 8 weeks
  Clinical response for platelets was assessed as the number of participants achieving a hematological improvement - platelets (HI-P). Participants will be characterized and stratified as platelets < or ≥ 20 x 10^9/L, with response defined as follows.
  * < 20 x 10^9/L = increase in platelets from < 20 x 10^9/L to > 20 x 10^9/L AND by ≥ 100%
  * ≥ 20 x 10^9/L = absolute increase in platelets of 30 x 10^9/L The outcome will be reported as the number of participants that achieve the response, a number without dispersion.
Clinical Response: Hematological Improvement - Neutrophils (HI-N) | 8 weeks
  Clinical response for neutrophils was assessed as the number of participants achieving a hematological improvement - neutrophils (HI-N). Response defined as an absolute increase in neutrophils > 0.5 x 10^9/L that is also an increase of ≥ 100%.
  The outcome will be reported as the number of participants that achieve the response, a number without dispersion.
Red Blood Cell (RBC) transfusion independence (RBC TI) | 12 months
  Clinical response for red blood cells was assessed as the number of participants who were transfusion dependent that achieve red blood cell (RBC) transfusion independence (RBC TI) for for 8 weeks or longer. The outcome will be reported as the number of participants that achieve the response, a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Tian Yi Zhang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Institute, Palo Alto, California, United States